CLINICAL TRIAL: NCT05369481
Title: Comparative Study Between the Efficacy of Topical Sildenafil 2% and Topical Minoxidil 5% in the Treatment of Male Androgenic Alopecia
Brief Title: Comparison Between Efficacy of Topical Sildenafil 2% and Topical Minoxidil 5% in Treatment of Androgenic Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohammed Abd El Mawgoud Amer (Other)
Responsible Party: Sponsor-Investigator, Mohammed Abd El Mawgoud Amer, Professor, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Male Androgenic Alopecia
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildenafil 2% (Experimental): will receive topical sildenafil 2% twice daily for 6 months.
  Interventions: Drug: Sildenafil 2%
- Minoxidil 5 % (Experimental): will receive topical minoxidil 5 % twice daily for 6 months
  Interventions: Drug: Minoxidil 5 %

INTERVENTIONS:
Drug: Sildenafil 2% — Patients with male androgenic alopecia will be given topical Sildenafil 2% to apply twice daily for 6 consecutive months and then follow up.
  Other Names: Local Scalp Injection
  Arms: Sildenafil 2%
Drug: Minoxidil 5 % — Patients with male androgenic alopecia will be given topical Minoxidil 5 % to apply twice daily for 6 consecutive months and then follow up.
  Other Names: Local Scalp Injection
  Arms: Minoxidil 5 %

SUMMARY:
Androgenetic alopecia (AGA) is hair loss with specific clinical pattern, It Is characterized by follicular miniaturization, which occurs due to systemic androgens and genetic factors. Prevalence differs according to ethnic groups. It is more common and more severe in white men than in Asian and black men. The incidence increases with age. According to Hamilton's study, the prevalence is 30% in men at the age of 30, and 50% in the age of 50. Generally, the age of onset is the 3rd and 4th decade.

DETAILED DESCRIPTION:
Androgenetic alopecia may affect self-esteem and quality of life in several affected individuals. There are two FDA-approved drugs for pattern baldness: topical minoxidil and finasteride, both of which require at least a 4- to 6-month trial before noticing improvement and must be used indefinitely to maintain a response. As such, medication adherence often can be poor. Furthermore, initiation of the drug may cause an initial shedding phase.

Minoxidil was the first and, so far, the only topical product that has been FDA approved for the treatment of AGA. Minoxidil was originally developed as an oral medication for hypertension. Hypertrichosis was found in 24-100 % of patients treated with oral minoxidil, which led to the treatment of AGA with topical minoxidil.

Androgenic Alopecia is caused by the overproduction of 5αdihydrotestosterone (5α-DHT), a potent androgen within the hair follicle, specifically the dermal papilla (DP) cells that are the main regulators of hair growth and are the only site of 5α-DHT action.

Sildenafil is a selective inhibitor of phosphodiesterase 5 and was originally developed as an anti-anginal drug due to its vasodilatory and antiplatelet coagulation properties. Sildenafil enhances the proliferation of human dermal papilla cells and up-regulates the mRNA expression of vascular endothelial growth factor and platelet-derived growth factor (PDGF) which are responsible for hair growth.

Topical sildenafil 1% has been used in the treatment of male androgenic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects clinically and dermoscopic diagnosed with AGA.
* Age ranges from 18 to 45 years old.
* Males
* Willingness to provide pictures and follow-up studies.

Exclusion Criteria:

* Patients who received any topical or systemic treatment for AGA during the last 6 months,
* Patients who had other types of alopecia such as alopecia areata, alopecia totalis, telogen effluvium, anagen effluvium, and acquired cicatricial alopecia.
* Patients with anemia, thyroid disease, and vitamin D deficiency,
* Any autoimmune disease or chronic debilitating disease (chronic renal failure, congestive heart failure, hepatic patients, cancer patients).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Improvement changes | 6 months
  improvement will be assessed by comparing the trichoscopic photos before and after treatment as regard hair density

SECONDARY OUTCOMES:
Patient's satisfaction | 6 months
  by asking the patients and changes in dermatology life Quality Index score as it reflects the quality of life related to skin manifestations
Complications | 6 months
  infection and bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Amer, MD, Principal Investigator — Al-Azhar university Hospital
Locations (1):
- AL-Azhar University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No